CLINICAL TRIAL: NCT02266186
Title: Treatment of Severe Fear of Childbirth With CBT, Comparison of ICBT With Traditional Live Therapy (Victoria)
Brief Title: Treatment of Severe Fear of Childbirth With CBT, Comparison of ICBT With Traditional Live Therapy
Acronym: (Victoria)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Klaas Wijma, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr2012/375-31
Record Dates: First submitted 2014-09-22; First posted 2014-10-16 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Tocophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Internet CBT (Experimental): Intervention:Internet-based cognitive behavioural therapy.
  Interventions: Behavioral: Internet based Cognitive behavioural therapy
- Traditional CBT (Active Comparator): Intervention:Traditional CBT given by a therapist following given modules.
  Interventions: Behavioral: Traditional Cognitive behavioural therapy
- Care as usual (No Intervention): Childbirth preparation according to local routine

INTERVENTIONS:
Behavioral: Traditional Cognitive behavioural therapy — Therapist supported live therapy
  Other Names: Traditional CBT .
  Arms: Traditional CBT
Behavioral: Internet based Cognitive behavioural therapy — Internetbased CBTwith limited therapist support
  Other Names: Internet CBT
  Arms: Internet CBT

SUMMARY:
The purpose of this project To study the efficacy of Internet-based guided self-help program of Cognitive Behaviour Therapy (ICBT) compared to traditional individual live CBT in a group of women with severe fear of childbirth (S-FOC). The treatment groups are compared with a control group receiving individual support at their antenatal clinics.

DETAILED DESCRIPTION:
In Sweden, every year, about 6000 pregnant women suffer from severe FOC with consequences for the women's psychological health before, during and after birth, the way they manage the childbirth, and for their postpartum mother-child interaction.

In this project we want to examine the effect of CBT on SFOC given in two different ways. We compare these results with a group receiving support given traditionally on the clinics. But also a group without S-FOC. In case there is a significant effect of CBT, that is comparable given live as well as ICBT, we should have developed an adequate way of treatment that could be implemented in ordinary health care.

Hypothesis: S-FOC decreases in same extent (30 units on the W-DEQ) in both of the treatment groups. The group with S-FOC,that gets treatment as usual is consuming more healthcare than the groups receiving therapy.

One hundred and twenty pregnant women with severe fear of childbirth (S-FOC) according to their sum score on the Wijma Expectancy/Experience Questionnaire (W-DEQ vers. A) ≥85, and 40 women without S-FOC (W-DEQ <85) are recruited at 7 participating clinics in Sweden. In a first baseline measuring phase 40 women with S-FOC and 40 women without S-FOC are followed as control groups, receiving, if necessary, treatment according to the local routine. In the intervention part of the study 80 women with S-FOC are randomized either into ICBT or live CBT.

1. ICBT is as effective as traditional live therapy.
2. ICBT is as efficient as traditional live therapy

   .
3. The effect will remain after the childbirth The successful therapy leads to

   * less fear after childbirth
   * less traumatic events during delivery
   * less cesareans or instrumental deliveries
   * less postpartum depressions
   * less appointments in urgency during pregnancy
   * better Mother-child relation at 3 months
   * better self-estimated quality of life

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in 16-30weeks of pregnancy at time for enrolment
* Able to read and write Swedish language
* having the possibility to use the internet during the therapy.

Exclusion Criteria:

* Suicidal, psychotic or schizophrenic symptoms.
* Not motivated to work with their fear.
* Ongoing psychological therapy because of fear of childbirth
* Non Swedish- speaking women

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Level of fear of childbirth | Change baseline to after 8 weeks of treatment
  self rating with: Wijma Expectancy/Experience Questionnaire version A (W-DEQ vers. A)

SECONDARY OUTCOMES:
Level of trauma | Change from baseline to 3 months after delivery
  self rating with: Traumatic Event Scale (TES)
Level of anxiety and depression | Change from baseline to 3 months after delivery
  self rating with: Hospital anxiety and depression scale (HADS)

OTHER OUTCOMES:
Number of women delivered vaginally | 3 months after delivery
  Number of women delivered vaginally
  Influence of fear of childbirth on mother-child interaction ( self rating with MAMA) Self estimated quality of life EQ5D
Appointments | 3 months after delivery
  Appointments during pregnancy at Obstetrical department
Sick leave | 3 months after delivery
  Number of women at Sick leave during pregnancy
Mother-child interaction postpartum | 3 months after delivery
  Self-estimated with MAMA
Self-estimated quality of life | 3 moths after delivery
  Self-estimated with EQ5D

CONTACTS AND LOCATIONS:
Overall Officials: Klaas WIjma, Professor, Study Director — Linkoeping University
Locations (1):
- Kvinnokliniken, Vrinnevisjukhuset, Norrköping, Sweden

REFERENCES:
- See also: Homepage — https://www.iterapi.se/sites/victoria/